CLINICAL TRIAL: NCT02629159
Title: A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) to Placebo and to Adalimumab in Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Are on a Stable Background of Methotrexate (MTX) and Who Have an Inadequate Response to MTX (MTX-IR)
Brief Title: A Study Comparing Upadacitinib (ABT-494) to Placebo and to Adalimumab in Adults With Rheumatoid Arthritis Who Are on a Stable Dose of Methotrexate and Who Have an Inadequate Response to Methotrexate
Acronym: SELECT-COMPARE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-465; 2022-501017-31-00 (Other: EU CT)
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal disease; Arthritis; Joint disease; Anti-inflammatory agents; Antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — Adalimumab; upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo followed by ABT-494 (Placebo Comparator): Participants were to receive placebo to upadacitinib orally once daily (QD) and placebo to adalimumab by subcutaneous injection once every two weeks (eow) for up to 26 weeks. Participants who did not achieve a ≥ 20% improvement in tender joint count (TJC) and swollen joint count (SJC) at Weeks 14, 18, or 22 compared to Baseline were to be switched to 15 mg upadacitinib orally QD. At Week 26, all remaining participants were to be switched to 15 mg upadacitinib QD until Week 48 (end of Period 1).
  Participants who complete Period 1 will continue to receive 15 mg upadacitinib orally QD for up to 5 years in Period 2.
  Interventions: Drug: Placebo for Adalimumab; Drug: Placebo for Upadacitinib; Drug: Upadacitinib
- Adalimumab (Active Comparator): Participants were to receive placebo to upadacitinib orally QD and 40 mg adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were to be switched to 15 mg upadacitinib orally QD. At Week 26 remaining participants who did not achieve low disease activity (defined as Clinical Disease Activity Index [CDAI] ≤ 10) were to be switched to 15 mg upadacitinib orally QD until Week 48.
  Participants who complete Period 1 will continue to receive the same treatment assigned at the end of Period 1 (15 mg upadacitinib QD or 40 mg adalimumab eow) for up to 5 years in Period 2.
  Interventions: Drug: Adalimumab; Drug: Placebo for Upadacitinib; Drug: Upadacitinib
- Upadacitinib (Experimental): Participants were to receive 15 mg upadacitinib orally QD and placebo to adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were to be switched to 40 mg adalimumab eow. At Week 26 remaining participants who did not achieve low disease activity (defined as CDAI ≤ 10) were to be switched to 40 mg adalimumab eow until Week 48.
  Participants who complete Period 1 will continue to receive the same treatment assigned at the end of Period 1 (15 mg upadacitinib QD or 40 mg adalimumab eow) for up to 5 years in Period 2.
  Interventions: Drug: Placebo for Adalimumab; Drug: Adalimumab; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo for Adalimumab — Administered by subcutaneous injection once every other week
  Arms: Placebo followed by ABT-494; Upadacitinib
Drug: Adalimumab — Administered by subcutaneous injection once every other week
  Other Names: Humira
  Arms: Adalimumab; Upadacitinib
Drug: Placebo for Upadacitinib — Tablets taken orally once a day
  Arms: Adalimumab; Placebo followed by ABT-494
Drug: Upadacitinib — Tablets taken orally once a day
  Other Names: ABT-494

SUMMARY:
The purpose of this study was to assess efficacy, including inhibition of radiographic progression, and safety with upadacitinib versus placebo and versus an active comparator, adalimumab, in adults with with moderately to severely active rheumatoid arthritis (RA) who are on a stable background of methotrexate (MTX and who have an inadequate response to MTX.

DETAILED DESCRIPTION:
This study consists of a 48-week double-blind treatment period (Period 1) and a long-term extension period (Period 2).

Period 1 is a 48-week randomized, double-blind, parallel-group, placebo-controlled and active comparator-controlled period designed to compare the safety and efficacy of upadacitinib versus placebo, and versus adalimumab. Participants will be randomized in a 2:2:1 ratio to one of three treatment groups:

* Placebo (up to Week 26)
* Upadacitinib 15 mg once daily (QD)
* Adalimumab 40 mg every other week (eow)

Participants randomized to placebo who do not achieve a ≥ 20% improvement in tender joint count (TJC) and swollen joint count (SJC) at Weeks 14, 18, or 22 compared to Baseline will be switched to blinded upadacitinib treatment. At Week 26, all participants still receiving placebo will be switched to blinded upadacitinib treatment regardless of clinical response.

Participants randomized to adalimumab who do not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline will be switched to blinded upadacitinib. Participants still receiving adalimumab at Week 26 who do not achieve low disease activity (LDA) according to Clinical Disease Activity Index (CDAI; LDA is defined as CDAI ≤ 10) will be switched to blinded upadacitinib treatment to Week 48.

Participants randomized to upadacitinib who do not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline will be switched to blinded adalimumab; participants still receiving upadacitinib at Week 26 who do not achieve LDA (CDAI ≤ 10) will be switched to blinded adalimumab treatment to Week 48.

Participants who complete the Week 48 visit (end of Period 1) will enter the long-term extension phase of the study (Period 2), for up to 5 years. Participants will continue study treatment as assigned at the end of Period 1. Starting at the Week 48 and thereafter, at least 20% improvement in both TJC and SJC compared to Baseline is required to remain on study drug. Anyone who does not fulfill this criterion at 2 consecutive visits (starting at Week 48) will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, at least 18 years old.
* Diagnosis of RA for greater than or equal to 3 months.
* Subjects must have been on oral or parenteral methotrexate (MTX) therapy greater than or equal to 3 months and on a stable prescription of greater than or equal to 15 to 25 mg/week (or greater than or equal to 10 mg/week in subjects intolerant of MTX at doses greater than or equal to 12.5 mg/week) for at least 4 weeks prior to the first dose of study drug. In addition all subjects should take a dietary supplement of folic acid or folinic acid throughout the study participation.
* Meets the following minimum disease activity criteria: greater than or equal to 6 swollen joints (based on 66 joint counts) and greater than or equal to 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.
* At least one of the following at Screening: greater than or equal to 3 bone erosions on x-ray OR greater than or equal to 1 bone erosion and a positive rheumatoid factor OR greater than or equal to 1 bone erosion and a positive anti-cyclic citrullinated peptide autoantibodies.
* Subjects with prior exposure to only one biological disease-modifying anti-rheumatic drugs (bDMARD) (except adalimumab) may be enrolled (up to 20% of total study population) if they have documented evidence of intolerance to the bDMARD or limited exposure (less than 3 months), but required washout periods need to be satisfied.
* Except for MTX, subject must have discontinued all conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs).

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Subjects who have been exposed to adalimumab or who are considered inadequate responders to bDMARD therapy as determined by the Investigator.
* History of inflammatory joint disease other than RA. History of secondary Sjogren's Syndrome is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1629 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2027-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (370):
- United States (109):
  - Achieve Clinical Research, LLC /ID# 143136, Birmingham, Alabama
  - AZ Arthritis and Rheum Assoc /ID# 143130, Mesa, Arizona
  - SunValley Arthritis Center, Lt /ID# 143123, Peoria, Arizona
  - Elite Clinical Studies, LLC /ID# 144881, Phoenix, Arizona
  - AZ Arthritis and Rheum Researc /ID# 143080, Phoenix, Arizona
  - AZ Arthritis and Rheum Researc /ID# 143121, Phoenix, Arizona
  - AZ Arthritis & Rheuma Research /ID# 143131, Phoenix, Arizona
  - Arizona Research Center, Inc. /ID# 144877, Phoenix, Arizona
  - AZ Arthritis & Rheum Research /ID# 156093, Sun City, Arizona
  - University of Arizona Cancer Center - North Campus /ID# 143114, Tucson, Arizona
  - Osteoporosis Medical Center /ID# 153935, Beverly Hills, California
  - T. Joseph Raoof, MD, Inc. /ID# 144884, Encino, California
  - Rheumatology Ctr of San Diego /ID# 153747, Escondido, California
  - C.V. Mehta MD, Med Corporation /ID# 143116, Hemet, California
  - Allergy and Rheum Med Clin /ID# 146083, La Jolla, California
  - Kotha and Kotha /ID# 161046, La Mesa, California
  - TriWest Research Associates- La Mesa /ID# 143115, La Mesa, California
  - Valerius Med Grp & Res Ctr /ID# 143120, Los Alamitos, California
  - Discovery MM Services, Inc /ID# 163504, Los Angeles, California
  - Desert Medical Advances /ID# 143097, Palm Desert, California
  - Sierra Rheumatology /ID# 155672, Roseville, California
  - Robin K. Dore MD, Inc /ID# 143090, Tustin, California
  - Medvin Clinical Research /ID# 148362, Whittier, California
  - Arthritis Assoc & Osteo Ctr /ID# 143122, Colorado Springs, Colorado
  - Arthritis and Rheum Clin N. CO /ID# 156094, Fort Collins, Colorado
  - AARDS Research, Inc. /ID# 154190, Aventura, Florida
  - ZASA Clinical Research /ID# 143134, Boynton Beach, Florida
  - Clinical Res of West FL, Inc. /ID# 143112, Clearwater, Florida
  - International Medical Research /ID# 143132, Daytona Beach, Florida
  - Lakes Research, LLC /ID# 145630, Miami, Florida
  - FL Med Ctr and Research, Inc. /ID# 143081, Miami, Florida
  - Ctr Arthritis & Rheumatic Dise /ID# 143135, Miami, Florida
  - Precision Research Org, LLC /ID# 143092, Miami Lakes, Florida
  - Advanced Clin Res of Orlando /ID# 154617, Ocoee, Florida
  - Rheum Assoc of Central FL /ID# 145632, Orlando, Florida
  - Omega Research Consultants /ID# 145635, Orlando, Florida
  - HMD Research LLC /ID# 163292, Orlando, Florida
  - Arthritis Research of Florida /ID# 143125, Palm Harbor, Florida
  - Arthritis Center, Inc. /ID# 145647, Palm Harbor, Florida
  - St. Anthony Comprehsve Res Ins /ID# 143095, St. Petersburg, Florida
  - Clinical Research West FL /ID# 148358, Tampa, Florida
  - SW FL Clin Res Ctr, Tampa, FL /ID# 143117, Tampa, Florida
  - BayCare Medical Group, Inc. /ID# 143085, Tampa, Florida
  - Lovelace Scientific Resources /ID# 143106, Venice, Florida
  - Arthritis and Rheumatology /ID# 155668, Atlanta, Georgia
  - Arthritis Center of North GA /ID# 155258, Gainesville, Georgia
  - North Georgia Rheumatology Grp /ID# 147170, Lawrenceville, Georgia
  - Advanced Clinical Research /ID# 153090, Meridian, Idaho
  - Great Lakes Clinical Trials /ID# 148357, Chicago, Illinois
  - Arthritis Treatment Center /ID# 155260, Frederick, Maryland
  - The Center for Rheumatology & /ID# 151356, Wheaton, Maryland
  - Clinical Pharmacology Study Gr /ID# 143082, Worcester, Massachusetts
  - Advanced Rheumatology, PC /ID# 143118, Lansing, Michigan
  - Shores Rheumatology, PC /ID# 162977, Saint Clair Shores, Michigan
  - St. Luke's Hospital /ID# 156750, Duluth, Minnesota
  - North Mississippi Med Clinics /ID# 145636, Tupelo, Mississippi
  - Physician Res. Collaboration /ID# 143087, Lincoln, Nebraska
  - Quality Clinical Research Inc. /ID# 156394, Omaha, Nebraska
  - Atlantic Coast Research /ID# 148355, Toms River, New Jersey
  - Ocean Rheumatology, PA /ID# 143111, Toms River, New Jersey
  - Arthritis Rheumatic Back Disorder /ID# 143102, Voorhees Township, New Jersey
  - Albuquerque Clinical Trials, Inc /ID# 143083, Albuquerque, New Mexico
  - Arthritis and Osteo Assoc /ID# 143127, Las Cruces, New Mexico
  - St. Lawrence Health System /ID# 161619, Potsdam, New York
  - Joint & Muscle Research Instit /ID# 143119, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 143101, Charlotte, North Carolina
  - EmergeOrtho, P.A. /ID# 143100, Durham, North Carolina
  - Cape Fear Arthritis Care /ID# 148361, Leland, North Carolina
  - Coastal Carolina Health Care /ID# 148359, New Bern, North Carolina
  - Shanahan Rheuma & Immuno /ID# 145643, Raleigh, North Carolina
  - Clinical Research Solutions, LLC /ID# 154619, Dayton, Ohio
  - Arthritis Assoc of NW Ohio /ID# 143094, Toledo, Ohio
  - Healthcare Research Consultant /ID# 143129, Tulsa, Oklahoma
  - Altoona Ctr Clinical Res /ID# 143110, Duncansville, Pennsylvania
  - Clinical Research Ctr Reading /ID# 143133, Wyomissing, Pennsylvania
  - Columbia Arthritis Center /ID# 153730, Columbia, South Carolina
  - Innovative Clinical Research /ID# 145637, Greenville, South Carolina
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 143091, Summerville, South Carolina
  - Arthritis Associates, PLLC /ID# 155490, Kingsport, Tennessee
  - Rheumatology Consultants, PLLC /ID# 153731, Knoxville, Tennessee
  - Dr. Ramesh Gupta /ID# 143099, Memphis, Tennessee
  - Austin Regional Clinic /ID# 143084, Austin, Texas
  - Diagnostic Group Integrated He /ID# 148356, Beaumont, Texas
  - Arthritis Care and Diagnostic /ID# 150677, Dallas, Texas
  - Metroplex Clinical Research /ID# 145631, Dallas, Texas
  - Doctor's Hosp at Renaissance /ID# 154616, Edinburg, Texas
  - MedResearch Inc. /ID# 154618, El Paso, Texas
  - Accurate Clinical Management /ID# 145644, Houston, Texas
  - Accurate Clinical Research /ID# 145645, Houston, Texas
  - Rheumatology Clinic of Houston /ID# 150921, Houston, Texas
  - Houston Institute for Clin Res /ID# 144879, Houston, Texas
  - Pioneer Research Solutions, Inc. /ID# 145640, Houston, Texas
  - Arthritis Consultants, P.A. /ID# 144880, Killeen, Texas
  - Arthritis & Osteoporosis Assoc /ID# 147364, Lubbock, Texas
  - P&I Clinical Research /ID# 161625, Lufkin, Texas
  - SW Rheumatology Res. LLC /ID# 143126, Mesquite, Texas
  - Discovery MM Services, Inc. /ID# 162578, Missouri City, Texas
  - Discovery MM Services, Inc. /ID# 163183, Missouri City, Texas
  - Discovery MM Services, Inc. /ID# 163184, Missouri City, Texas
  - Sun Research Institute /ID# 159539, San Antonio, Texas
  - Accurate Clinical Management /ID# 143089, San Antonio, Texas
  - Arthritis & Osteo Ctr of S. TX /ID# 143103, San Antonio, Texas
  - DM Clinical Research /ID# 151357, Tomball, Texas
  - Arthritis Clinic of N. VA, P.C /ID# 143109, Arlington, Virginia
  - Ctr for Arth and Rheum Disease /ID# 143113, Chesapeake, Virginia
  - Arthritis Northwest, PLLC /ID# 143088, Spokane, Washington
  - The Vancouver Clinic, INC. PS /ID# 143107, Vancouver, Washington
  - West Virginia Research Inst /ID# 153088, South Charleston, West Virginia
  - Rheumatology and Immunotherapy Center /ID# 145646, Franklin, Wisconsin
- Argentina (14):
  - Aprillus Asistencia e Investig /ID# 148406, Capital Federal, Buenos Aires
  - Mautalen Salud e Investigacion /ID# 142843, Buenos Aires
  - Fundacion Sanatorio Guemes /ID# 148405, Buenos Aires
  - Consultorio Reumatologic Pampa /ID# 144853, Buenos Aires
  - Cemic /Id# 148404, Buenos Aires
  - Org Medica de Investigacion /ID# 144855, Buenos Aires
  - Inst. Rheumatologic Strusberg /ID# 145601, Córdoba
  - Consultora Integral de Salud S /ID# 144856, Córdoba
  - Instituto CAICI /ID# 144854, Rosario, Santa FE
  - Cordis S.A. /Id# 152622, Salta
  - Iari /Id# 151293, San Fernando
  - Centro Integral de Reumatologi /ID# 142845, San Miguel de Tucumán
  - Centro Medico Privado/Reuma /ID# 142842, San Miguel de Tucumán
  - Centro de Enfermedades /ID# 153542, Santa Fe
- Australia (2):
  - Royal Prince Alfred Hospital /ID# 144857, Camperdown, New South Wales
  - Emeritus Research /ID# 142848, Camberwell, Victoria
- LKH-Univ. Klinikum Graz /ID# 142851, Graz, Austria
- First City Clinical Hospital /ID# 158011, Minsk, Belarus
- Belgium (5):
  - Cliniques Universitaires Saint Luc /ID# 142858, Woluwe-Saint-Lambert, Brussels Capital
  - Rhumaconsult SPRL /ID# 142860, Charleroi, Hainaut
  - CHU de Liege /ID# 148401, Liège, Liege
  - UZ Gent /ID# 142859, Ghent, Oost-Vlaanderen
  - CHU Ambroise Pare /ID# 152953, Mons
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska /ID# 142862, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 142863, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 142865, Sarajevo
- Brazil (7):
  - CIP - Centro Internacional de Pesquisa /ID# 142872, Goiânia, Goiás
  - Hc Ufmg /Id# 142868, Belo Horizonte, Minas Gerais
  - Ceti - Centro de Estudos Em Terapias Inovadoras Ltda /Id# 142871, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 142870, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 142869, Porto Alegre, Rio Grande do Sul
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos Ltda /ID# 142867, São Paulo, São Paulo
  - CCBR Brasil /ID# 150918, Rio de Janeiro
- Bulgaria (5):
  - MHAT Trimontsium /ID# 142874, Plovdiv
  - UMHAT Pulmed OOD /ID# 142877, Plovdiv
  - MHAT Kaspela /ID# 142873, Plovdiv
  - Diagnostic Consultative Center /ID# 142875, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 142876, Sofia
- Canada (6):
  - Manitoba Clinic /ID# 161434, Winnipeg, Manitoba
  - Ciads /Id# 142880, Winnipeg, Manitoba
  - St. Clare's Mercy Hospital /ID# 142879, St. John's, Newfoundland and Labrador
  - Adachi Medicine Prof. Corp /ID# 154205, Hamilton, Ontario
  - CA Ctr for Clin Trials CCCT /ID# 157379, Thornhill, Ontario
  - Groupe de Recherche en Maladies Osseuses /ID# 142878, Sainte-Foy, Quebec
- Chile (12):
  - Ctr de Inv Clinica del Sur /ID# 142888, Temuco, Región de la Araucanía
  - Reg. Clinical Hosptial Concepcion /ID# 151271, Concepción
  - Corp de Beneficencia Osorno /ID# 147941, Osorno
  - Someal /Id# 144704, Providencia-santiago
  - Quantum Research LTDA. /ID# 142893, Puerto Varas
  - Quantum Research Stgo. /ID# 157933, Santiago
  - Soc. de Prestaciones medicas y Paramedicas Goecke /ID# 142890, Santiago
  - Clinica DermaCross /ID# 142892, Santiago
  - Investigaciones Medicas SSMSO /ID# 151686, Santiago
  - Centro Inter Estud Clin CIEC /ID# 144777, Santiago
  - Centro Medico de Reumatologia /ID# 148402, Temuco
  - Cinvec /Id# 144705, Viña del Mar
- Colombia (6):
  - Centro de Investigacion en Reumatologia y Especialidades Medicas- CIREEM SAS /ID# 142898, Bogota, Cundinamarca
  - Ctr Int de Reum del Caribe SAS /ID# 142894, Barranquilla
  - Fund Inst de Reum F. Chalem /ID# 149847, Bogota DC
  - Riesgo de Fractura S.A - CAYRE /ID# 142896, Bogotá
  - Medicity S.A.S. /ID# 144860, Bucaramanga
  - Centro Integral de Reumatologi /ID# 142897, Medellín
- Croatia (5):
  - Klinicki bolnicki centar Rijeka /ID# 160232, Rijeka, Primorje-Gorski Kotar County
  - Klinicki bolnicki centar Split /ID# 152530, Split
  - Clinical Hospital Dubrava /ID# 142900, Zagreb
  - Medical Center Kuna-Peric /ID# 142901, Zagreb
  - Poliklinika Bonifarm /ID# 142899, Zagreb
- Czechia (11):
  - L.K.N. Arthrocentrum, s.r.o /ID# 145961, Hlučín, Moravskoslezský kraj
  - CTCenter MaVe, s.r.o. /ID# 142905, Olomouc, Olomoucký kraj
  - Revmatologicky ustav Praha /ID# 142904, Prague, Praha 2
  - Nuselská poliklinika, Revmatologie /ID# 144862, Prague, Praha 4
  - Revmatologická ambulance /ID# 145963, Prague, Praha 4
  - Thomayerova nemocnice /ID# 145962, Prague, Praha 4
  - REVMACLINIC s.r.o. /ID# 142906, Brno
  - Revmatologie Bruntal, s.r.o /ID# 142903, Bruntál
  - Revmatologicka a interni ambul /ID# 142907, Kladno
  - Revmatologie MUDr. Klara Sirov /ID# 142908, Ostrava
  - Arthromed, s.r.o. /ID# 144706, Pardubice
- Denmark (2):
  - Aarhus University Hospital /ID# 158838, Aarhus N, Central Jutland
  - Regionhospital Silkeborg /ID# 142914, Silkeborg
- Estonia (5):
  - Center of Clinical and Basic Research /ID# 142922, Tallinn, Harju
  - MediTrials /ID# 151870, Tartu, Tartu
  - Paernu Hospital /ID# 142921, Pärnu
  - East Tallinn Central Hospital /ID# 142923, Tallinn
  - North Estonian Medical Centre /ID# 145454, Tallinn
- France (10):
  - Hopital Universitaire Purpan /ID# 144707, Toulouse, Haute-Garonne
  - CHRU Lille - Hôpital Claude Huriez /ID# 151312, Lille, Hauts-de-France
  - Hopital Saint Eloi /ID# 142925, Montpellier, Herault
  - CHU Bordeaux-Hopital Pellegrin /ID# 145618, Bordeaux
  - Hopital de la Cote de Nacre /ID# 145616, Caen
  - CHU Gabriel Montpied /ID# 145619, Clermont-Ferrand
  - Hopital de la Conception /ID# 142926, Marseille
  - Hopital Pitie Salpetriere /ID# 145605, Paris
  - CHU de Rennes - Hospital Sud /ID# 151957, Rennes
  - CHU Strasbourg Hautepierre Hos /ID# 144708, Strasbourg
- Germany (6):
  - Uniklinik Koln /ID# 145964, Cologne, North Rhine-Westphalia
  - Rheumazentrum Ruhrgebiet /ID# 145620, Herne, North Rhine-Westphalia
  - Praxis Walter, Rendsburg /ID# 142932, Rendsburg, Schleswig-Holstein
  - Med Versorgungszentrum AGILOME /ID# 154975, Chemnitz
  - Rheumaforschungszentrum II /ID# 142930, Hamburg
  - LMU Klinikum der Universität München /ID# 142931, Munich
- Greece (3):
  - General Hospital of Athens Laiko /ID# 142934, Athens, Attica
  - University General Hospital Attikon /ID# 142933, Athens, Attica
  - General Hospital of Athens Ippokratio /ID# 142935, Athens
- Hong Kong (2):
  - Queen Mary Hospital /ID# 142938, Hong Kong
  - Tuen Mun Hospital /ID# 142939, Tuenmen
- Hungary (11):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 142951, Miskolc, Borsod-Abauj Zemplen county
  - Qualiclinic Kft. /ID# 142953, Budapest III, Pest County
  - Markusovszky Egyetemi Oktatókórház /ID# 145621, Szombathely, Vas County
  - Vital Medical Center Orvosi es /ID# 145950, Veszprém, Veszprém megye
  - Budai Irgalmasrendi Korhaz /ID# 142952, Budapest
  - Revita Reumatologiai Rendelo /ID# 142950, Budapest
  - Synexus Magyarorszag Kft. /ID# 153061, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 142948, Debrecen
  - Hevizgyogyfurdo es Szent Andra /ID# 142949, Hévíz
  - Kiskunhalasi Semmelweis Korhaz /ID# 151944, Kiskunhalas
  - Pest Megyei Flor Ferenc Korhaz /ID# 142954, Kistarcsa
- St Vincent's University Hosp /ID# 142957, Dublin, Ireland
- Israel (5):
  - Tel Aviv Sourasky Medical Ctr /ID# 144709, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 152050, Haifa
  - Bnai Zion Medical Center /ID# 151958, Haifa
  - The Lady Davis Carmel MC /ID# 142960, Haifa
  - Sheba Medical Center /ID# 145965, Ramat Gan
- Italy (4):
  - Istituto Clinico Humanitas /ID# 147528, Rozzano, Milano
  - AOU Citta della Salute Scienza /ID# 150070, Turin, Piedmont
  - Azienda Ospedaliera Luigi Sacc /ID# 142966, Milan
  - A.O.U.I. di Verona Policlinico /ID# 142963, Verona
- Kazakhstan (4):
  - JSC Nat Scientific Med Res Ctr /ID# 142971, Astana
  - Karaganda State Medical Univ /ID# 153433, Karaganda
  - Semey State Medical University /ID# 152659, Semey
  - Regional Clinical Hospital /ID# 147168, Shymkent
- Latvia (5):
  - LTD M+M Centers /ID# 142984, Ādaži
  - Daugavpils Regional Hospital /ID# 142982, Daugavpils
  - D.Saulites-Kandevicas PP /ID# 142985, Liepāja
  - Clinic ORTO /ID# 142983, Riga
  - Riga East Clinical Univ Hosp /ID# 142981, Riga
- Lithuania (2):
  - Hosp Lithuanian Univ Health Sc /ID# 142986, Kaunas, Kaunas County
  - Vilnius University Hospital /ID# 142987, Vilnius
- Malaysia (5):
  - Hospital Raja Perempuan Zainab II /ID# 157862, Kota Bharu, Kelantan
  - Hospital Selayang /ID# 156756, Batu Caves
  - Hospital Umum Sarawak /ID# 142990, Kuching
  - Hospital Putrajaya /ID# 142989, Putrajaya
  - Hospital Tuanku Ja afar /ID# 142988, Seremban
- Mexico (6):
  - Clinstile, S.A. de C.V. /ID# 144866, Cuauhtémoc, Mexico City
  - Hosp. Univ. Dr. Jose E. Gonz /ID# 142992, Monterrey, Nuevo León
  - Invest y Biomed de Chihuahua /ID# 142996, Chihuahua City
  - RM Pharma Specialists, S.A de C.V /ID# 142994, Mexico City
  - Hospital de Jesús Nazareno /ID# 142993, Mexico City
  - Centro Peninsular de Investiga /ID# 148159, Mérida
- New Zealand (3):
  - Waikato Hospital /ID# 143002, Hamilton, Waikato Region
  - Porter Rheumatology Ltd /ID# 143001, Nelson
  - Timaru Medical Specialists Ltd /ID# 143000, Timaru
- Poland (16):
  - NZOZ Nasz Lekarz /ID# 143004, Torun, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 152782, Krakow, Lesser Poland Voivodeship
  - Pratia MCM Krakow /ID# 143005, Krakow, Lesser Poland Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 145622, Wroclaw, Lower Silesian Voivodeship
  - REUMED Sp.z o.o. Filia nr 1 /ID# 148189, Lublin, Lublin Voivodeship
  - McBk Sc /Id# 143003, Grodzisk Mazowiecki, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie /ID# 151960, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED Warszawa Targowek /ID# 157621, Warsaw, Masovian Voivodeship
  - Osteo-Medic spolka cywilna /ID# 143006, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Sp. z o.o. Oddz. Poznan /ID# 163293, Gdynia, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddz. Poznan /ID# 163294, Gdynia, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddz. Poznan /ID# 163295, Gdynia, Pomeranian Voivodeship
  - Silmedic Sp z o.o /ID# 152914, Katowice, Silesian Voivodeship
  - ClinicMed Badurski i wspolnicy SJ /ID# 163300, Bialystok
  - Solumed Sp. zoo Cent Medyczne /ID# 152783, Poznan
  - Rheuma Medicus /ID# 143007, Warsaw
- Portugal (6):
  - Instituto Portugues De Reumatologia /ID# 148316, Lisbon, Lisbon District
  - Centro Hospitalar De Vila Nova /ID# 143010, Vila Nova de Gaia, Porto District
  - CCA Braga - Hospital de Braga /ID# 148317, Braga
  - Hospital CUF Descobertas /ID# 160539, Lisbon
  - Centro Hospitalar de Sao Joao, EPE /ID# 152871, Porto
  - Unidade Local De Saude Do Alto Minho /ID# 143009, Viana do Castelo
- Puerto Rico (2):
  - Ponce School of Medicine /ID# 151961, Ponce
  - GCM Medical Group /ID# 143011, San Juan
- Romania (7):
  - Spitalul Clinic Dr. I. Cantacuzino /ID# 143012, Bucharest, București
  - Spitalul Clinic Dr. I. Cantacuzino /ID# 143017, Bucharest, București
  - Spitalul Clinic Sf. Maria /ID# 144868, Bucharest
  - Spitalul Clinic Sf. Maria /ID# 144869, Bucharest
  - Spitalul Clinic Sf. Maria /ID# 145966, Bucharest
  - Spitalul Clinic de Recuperare /ID# 144867, Iași
  - Ecomed SRL /ID# 144870, Oradea
- Russia (17):
  - Family Outpatient clinic#4,LLC /ID# 148319, Korolev, Moscow
  - Clinical Hospital No.1 n.a. N.I.Pirogov /ID# 143138, Moscow, Moscow
  - Perm Clinical Center of FMBA /ID# 145627, Perm, Permskiy Kray
  - LLC Novaya Klinika /ID# 143019, Pyatigorsk, Stavropol Kray
  - Kazan State Medical University /ID# 144871, Kazan', Tatarstan, Respublika
  - Tver Regional Clinical Hosp. /ID# 143026, Tver', Tver Oblast
  - Сity Clinical Hospital #4 /ID# 143023, Ivanovo
  - Russian National Research Medi /ID# 143028, Moscow
  - City Clinical Hospital Botkina /ID# 145628, Moscow
  - Moscow State Univ Med and Dent /ID# 145623, Moscow
  - City Clinical Hospital #5 /ID# 148318, Nizhny Novgorod
  - Orenburg State Medical Academy /ID# 143018, Orenburg
  - Ryazan State Medical Universit /ID# 143031, Ryazan
  - II Dzhan Research Center /ID# 143027, Saint Petersburg
  - NW State Med Univ NA Mechnikov /ID# 143022, Saint Petersburg
  - Republican clinical hospital n /ID# 145626, Ufa
  - Ulyanovsk Regional Clin Hosp /ID# 143030, Ulyanovsk
- Serbia (6):
  - Institute for Rheumatology /ID# 143032, Belgrade, Beograd
  - Institute for Rheumatology /ID# 143035, Belgrade, Beograd
  - Institute for Rheumatology /ID# 143036, Belgrade, Beograd
  - Institute for Rheumatology /ID# 143037, Belgrade, Beograd
  - Special Hospital for Rheuma /ID# 143034, Novi Sad, Vojvodina
  - Clinical Center of Vojvodina /ID# 143033, Novi Sad, Vojvodina
- Slovakia (9):
  - MEDMAN s.r.o. /ID# 143045, Martin
  - Reumatologická ambulancia Reum.hapi s.r.o. /ID# 147169, Nové Mesto nad Váhom
  - REUMACENTRUM s.r.o. /ID# 143041, Partizánske
  - Slovak research center Team Member, Thermium s.r.o. /ID# 147614, Pieštany
  - Reumex, s.r.o. /ID# 143043, Rimavská Sobota
  - Reumatologicka ambulancia /ID# 144873, Sabinov
  - TIMMED spol. s r.o. /ID# 144872, Stará Lubovna
  - Reumatologicka ambulancia, LER /ID# 143044, Topoľčany
  - ALBAMED s.r.o. /ID# 143042, Zvolen
- South Africa (10):
  - Greenacres Hospital /ID# 144710, Port Elizabeth, Eastern Cape
  - Wits Clinical Research Site /ID# 148320, Johannesburg, Gauteng
  - University of Pretoria /ID# 148353, Pretoria, Gauteng
  - Jakaranda Hosp, Emmed Research /ID# 143046, Pretoria, Gauteng
  - Jakaranda Hosp, Emmed Research /ID# 145968, Pretoria, Gauteng
  - St. Augustine's Hospital /ID# 143047, Durban, KwaZulu-Natal
  - Synexus Helderberg Clinical Tr /ID# 148322, Cape Town, Western Cape
  - Arthritis Clinical Research Tr /ID# 144874, Cape Town, Western Cape
  - Tiervlei Trial Centre /ID# 153085, Cape Town, Western Cape
  - Winelands Medical Research Ctr /ID# 143048, Stellenbosch, Western Cape
- South Korea (9):
  - Kyungpook National Univ Hosp /ID# 162073, Daegu, Daegu Gwang Yeogsi
  - Chungnam National University Hospital /ID# 142977, Junggu, Daejeon Gwang Yeogsi
  - Inha University Hospital /ID# 150886, Junggu, Incheon Gwang Yeogsi
  - Chonnam National University Hospital /ID# 142975, Gwangju, Jeonranamdo
  - Hanyang University Seoul Hospi /ID# 142979, Seongdong-gu, Seoul Teugbyeolsi
  - Cath Univ Seoul St Mary's Hosp /ID# 142976, Seoul, Seoul Teugbyeolsi
  - Daegu Catholic University Med /ID# 142973, Daegu
  - Seoul National University Hospital /ID# 142978, Seoul
  - Asan Medical Center /ID# 142974, Seoul
- Spain (5):
  - H. Un. Marques de Valdecilla /ID# 143050, Santander, Cantabria
  - Comple Hosp Univ de A Coruna /ID# 143051, A Coruña
  - Hospital Universitario Reina S /ID# 153566, Córdoba
  - Clinica Gaias /ID# 143052, Santiago de Compostela
  - Complejo Hosp Santiago /ID# 153727, Santiago de Compostela
- Taiwan (8):
  - China Medical University Hosp /ID# 143058, Taichung, Taichung
  - National Taiwan Univ Hosp /ID# 143056, Taipei City, Taipei
  - Kaohsiung Medical University /ID# 143059, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital /ID# 143055, Kaohsiung City
  - Far Eastern Memorial Hospital /ID# 143061, New Taipei City
  - Chung Shan Medical University /ID# 143060, Taichung
  - Taipei Veterans General Hosp /ID# 157940, Taipei
  - Linkou Chang Gung Memorial Ho /ID# 143057, Taoyuan
- Turkey (Türkiye) (3):
  - Istanbul Universitesi Cerrahpa /ID# 156088, Cerrahpaşa
  - Istanbul Fizik Tedavi Rehabilitasyon Egitim ve Arastırma Hastanesi /ID# 143063, Istanbul
  - Izmir Katip Celebi Ataturk Training & Research Hospital /ID# 143062, Izmir
- Ukraine (8):
  - LLC Revmocentr /ID# 143067, Kiev, Kyiv Oblast
  - Lviv Regional Clinical Hospita /ID# 154450, Lviv, Lviv Oblast
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 143071, Vinnytsia, Vinnytsia Oblast
  - Regional Clinical Hospital /ID# 152025, Ivano-Frankivsk
  - NSC-Strazhesko Ist Cardiology /ID# 152030, Kiev
  - Lviv Municipal City Clinical /ID# 143068, Lviv
  - Odessa National Medical Univ /ID# 143072, Odesa
  - Zaporizhzhia Regional Clinical /ID# 143069, Zaporizhia
- United Kingdom (3):
  - The Royal Free Hospital /ID# 143074, London, London, City of
  - Queen Alexandra Hospital /ID# 143077, Portsmouth
  - Warrington + Halton Hosp NHS /ID# 143075, Warrington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Fleischmann R, Pangan AL, Song IH, Mysler E, Bessette L, Peterfy C, Durez P, Ostor AJ, Li Y, Zhou Y, Othman AA, Genovese MC. Upadacitinib Versus Placebo or Adalimumab in Patients With Rheumatoid Arthritis and an Inadequate Response to Methotrexate: Results of a Phase III, Double-Blind, Randomized Controlled Trial. Arthritis Rheumatol. 2019 Nov;71(11):1788-1800. doi: 10.1002/art.41032. Epub 2019 Aug 28. PMID 31287230
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Fleischmann R, Swierkot J, Penn SK, Durez P, Bessette L, Bu X, Khan N, Li Y, Peterfy CG, Tanaka Y, Mysler E. Long-term safety and efficacy of upadacitinib versus adalimumab in patients with rheumatoid arthritis: 5-year data from the phase 3, randomised SELECT-COMPARE study. RMD Open. 2024 May 28;10(2):e004007. doi: 10.1136/rmdopen-2023-004007. PMID 38806190
- [Derived] Fleischmann R, Blanco R, Van den Bosch F, Bessette L, Song Y, Penn SK, McDearmon-Blondell E, Khan N, Chan K, Mysler E. Long-term Efficacy and Safety Following Switch Between Upadacitinib and Adalimumab in Patients with Rheumatoid Arthritis: 5-Year Data from SELECT-COMPARE. Rheumatol Ther. 2024 Jun;11(3):599-615. doi: 10.1007/s40744-024-00658-1. Epub 2024 Mar 18. PMID 38498140
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Fleischmann R, Curtis JR, Charles-Schoeman C, Mysler E, Yamaoka K, Richez C, Palac H, Dilley D, Liu J, Strengholt S, Burmester G. Safety profile of upadacitinib in patients at risk of cardiovascular disease: integrated post hoc analysis of the SELECT phase III rheumatoid arthritis clinical programme. Ann Rheum Dis. 2023 Sep;82(9):1130-1141. doi: 10.1136/ard-2023-223916. Epub 2023 Jun 12. PMID 37308218
- [Derived] Conaghan PG, Pavelka K, Hsieh SC, Bonnington TL, Kent TC, Marchbank K, Edwards CJ. Evaluating the efficacy of upadacitinib in patients with moderate rheumatoid arthritis: a post-hoc analysis of the SELECT phase 3 trials. Rheumatol Adv Pract. 2023 Feb 8;7(1):rkad017. doi: 10.1093/rap/rkad017. eCollection 2023. PMID 36794283
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Kakehasi AM, Radominski SC, Baravalle MD, Palazuelos FCI, Garcia-Garcia C, Arruda MS, Curi M, Liu J, Qiao M, Velez-Sanchez P, Vargas JI. Safety of upadacitinib in Latin American patients with rheumatoid arthritis: an integrated safety analysis of the SELECT phase 3 clinical program. Clin Rheumatol. 2023 May;42(5):1249-1258. doi: 10.1007/s10067-023-06513-y. Epub 2023 Jan 30. PMID 36715850
- [Derived] Bergman M, Buch MH, Tanaka Y, Citera G, Bahlas S, Wong E, Song Y, Zueger P, Ali M, Strand V. Routine Assessment of Patient Index Data 3 (RAPID3) in Patients with Rheumatoid Arthritis Treated with Long-Term Upadacitinib Therapy in Five Randomized Controlled Trials. Rheumatol Ther. 2022 Dec;9(6):1517-1529. doi: 10.1007/s40744-022-00483-4. Epub 2022 Sep 20. PMID 36125701
- [Derived] Mysler E, Tanaka Y, Kavanaugh A, Aletaha D, Taylor PC, Song IH, Shaw T, Song Y, DeMasi R, Ali M, Fleischmann R. Impact of initial therapy with upadacitinib or adalimumab on achievement of 48-week treatment goals in patients with rheumatoid arthritis: post hoc analysis of SELECT-COMPARE. Rheumatology (Oxford). 2023 May 2;62(5):1804-1813. doi: 10.1093/rheumatology/keac477. PMID 36018230
- [Derived] Peterfy CG, Strand V, Friedman A, Hall S, Mysler E, Durez P, Baraliakos X, Enejosa JV, Shaw T, Li Y, Chen S, Song IH. Inhibition of structural joint damage progression with upadacitinib in rheumatoid arthritis: 1-year outcomes from the SELECT phase 3 program. Rheumatology (Oxford). 2022 Aug 3;61(8):3246-3256. doi: 10.1093/rheumatology/keab861. PMID 34897366
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Strand V, Tundia N, Bergman M, Ostor A, Durez P, Song IH, Enejosa J, Schlacher C, Song Y, Fleischmann R. Upadacitinib improves patient-reported outcomes vs placebo or adalimumab in patients with rheumatoid arthritis: results from SELECT-COMPARE. Rheumatology (Oxford). 2021 Dec 1;60(12):5583-5594. doi: 10.1093/rheumatology/keab158. PMID 33590829
- [Derived] Fleischmann RM, Blanco R, Hall S, Thomson GTD, Van den Bosch FE, Zerbini C, Bessette L, Enejosa J, Li Y, Song Y, DeMasi R, Song IH. Switching between Janus kinase inhibitor upadacitinib and adalimumab following insufficient response: efficacy and safety in patients with rheumatoid arthritis. Ann Rheum Dis. 2021 Apr;80(4):432-439. doi: 10.1136/annrheumdis-2020-218412. Epub 2020 Nov 4. PMID 33148701
- [Derived] Cohen SB, van Vollenhoven RF, Winthrop KL, Zerbini CAF, Tanaka Y, Bessette L, Zhang Y, Khan N, Hendrickson B, Enejosa JV, Burmester GR. Safety profile of upadacitinib in rheumatoid arthritis: integrated analysis from the SELECT phase III clinical programme. Ann Rheum Dis. 2021 Mar;80(3):304-311. doi: 10.1136/annrheumdis-2020-218510. Epub 2020 Oct 28. PMID 33115760
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- [Derived] Fleischmann RM, Genovese MC, Enejosa JV, Mysler E, Bessette L, Peterfy C, Durez P, Ostor A, Li Y, Song IH. Safety and effectiveness of upadacitinib or adalimumab plus methotrexate in patients with rheumatoid arthritis over 48 weeks with switch to alternate therapy in patients with insufficient response. Ann Rheum Dis. 2019 Nov;78(11):1454-1462. doi: 10.1136/annrheumdis-2019-215764. Epub 2019 Jul 30. PMID 31362993
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M14-465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active rheumatoid arthritis (RA) on a stable dose of methotrexate with an inadequate response were randomized at 286 study sites in 41 countries.
  This study is currently ongoing; results are reported as of the data cut-off date of 02 February 2018, when all participants were to have completed Week 26.
Pre-assignment Details: Participants were randomized in a 2:1:2 ratio to receive placebo, adalimumab, or upadacitinib. Randomization was stratified by prior exposure to biologic disease-modifying anti-rheumatic drug(s) (bDMARD) (yes/no) and geographic region.
  Rescue therapy was offered to participants who met protocol-specified criteria at Weeks 14, 18, 22, or 26.
Groups:
- Placebo: Participants randomized to receive placebo to upadacitinib orally once daily (QD) and placebo to adalimumab by subcutaneous injection once every two weeks (eow) for up to 26 weeks. Participants who did not achieve a ≥ 20% improvement in tender joint count (TJC) and swollen joint count (SJC) at Weeks 14, 18, or 22 compared to Baseline were switched to 15 mg upadacitinib orally QD. At Week 26, all remaining participants were switched to 15 mg upadacitinib QD.
- Adalimumab: Participants randomized to receive placebo to upadacitinib orally QD and 40 mg adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 15 mg upadacitinib orally QD. At Week 26 remaining participants who did not achieve low disease activity (defined as Clinical Disease Activity Index [CDAI] ≤ 10) were switched to 15 mg upadacitinib orally QD.
- Upadacitinib: Participants randomized to receive 15 mg upadacitinib orally QD and placebo to adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 40 mg adalimumab eow. At Week 26 remaining participants who did not achieve low disease activity (defined as CDAI ≤ 10) were switched to 40 mg adalimumab eow.
Period: Overall Study
Arm/Group | Placebo | Adalimumab | Upadacitinib
Started | 651 | 327 | 651
Received Assigned Study Drug | 651 | 327 | 650 (One participant received a placebo injection but no oral study drug before discontinuing the study)
Completed Week 14 on Study Drug | 620 | 300 | 620
Rescued at Week 14 | 231 | 56 | 78
Rescued at Week 18 | 48 (One participant rescued at week 18 did not receive any dose of upadacitinib) | 14 | 29
Rescued at Week 22 | 26 | 7 | 18
Completed (Participants who completed Week 26) | 595 | 288 | 600
Not Completed | 56 | 39 | 51
Not completed — Adverse Event | 17 | 20 | 22
Not completed — Withdrawal by Subject | 22 | 11 | 15
Not completed — Lost to Follow-up | 7 | 4 | 5
Not completed — Lack of Efficacy | 4 | 0 | 1
Not completed — Other | 6 | 4 | 8

BASELINE CHARACTERISTICS:
Population: The full analysis set consisted of all randomized participants who received at least 1 dose of study drug (placebo, adalimumab, or upadacitinib).
Groups:
- Placebo: Participants received placebo to upadacitinib orally once daily (QD) and placebo to adalimumab by subcutaneous injection once every two weeks (eow) for up to 26 weeks. Participants who did not achieve a ≥ 20% improvement in tender joint count (TJC) and swollen joint count (SJC) at Weeks 14, 18, or 22 compared to Baseline were switched to 15 mg upadacitinib orally QD.
- Adalimumab: Participants received placebo to upadacitinib orally QD and 40 mg adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 15 mg upadacitinib orally QD.
- Upadacitinib: Participants randomized to receive 15 mg upadacitinib orally QD and placebo to adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 40 mg adalimumab eow.
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab | Upadacitinib | Total
Number analyzed (Participants) | 651 | 327 | 651 | 1629
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (12.24) | 53.7 (11.70) | 54.2 (12.08) | 53.9 (12.07)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 91 | 39 | 81 | 211
  40 to 64 years | 437 | 232 | 439 | 1108
  ≥ 65 years | 123 | 56 | 131 | 310
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 512 | 259 | 521 | 1292
  Male | 139 | 68 | 130 | 337
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 206 | 106 | 215 | 527
  Not Hispanic or Latino | 445 | 221 | 436 | 1102
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 561 | 292 | 576 | 1429
  Black or African American | 38 | 17 | 33 | 88
  American Indian/Alaska Native | 2 | 1 | 1 | 4
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  Asian | 39 | 15 | 31 | 85
  Multiple | 10 | 2 | 10 | 22
Geographic Region [Count of Participants; unit: Participants]
  North America | 121 | 60 | 122 | 303
  South/Central America | 173 | 86 | 173 | 432
  Western Europe | 35 | 19 | 35 | 89
  Eastern Europe | 262 | 132 | 262 | 656
  Asia | 21 | 10 | 21 | 52
  Other | 39 | 20 | 38 | 97
Duration of Rheumatoid Arthritis Diagnosis [Mean (Standard Deviation); unit: years] | 8.3 (8.00) | 8.3 (8.41) | 8.1 (7.73) | 8.2 (7.97)
Tender Joint Count [Mean (Standard Deviation); unit: tender joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  tender joints | 26.0 (14.30) | 26.4 (15.16) | 26.4 (15.15) | 26.2 (14.81)
Swollen Joint Count [Mean (Standard Deviation); unit: swollen joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  swollen joints | 16.2 (8.97) | 16.3 (9.19) | 16.6 (10.31) | 16.4 (9.57)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain." Population: Participants with available data
  mm
    number analyzed (Participants) | 649 | 325 | 647 | 1621
    (all) | 65.0 (20.67) | 66.2 (20.51) | 65.7 (21.02) | 65.5 (20.77)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 649 | 324 | 647 | 1620
    (all) | 63.8 (21.49) | 65.8 (21.08) | 64.3 (21.83) | 64.4 (21.55)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100 mm, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 620 | 305 | 616 | 1541
    (all) | 66.0 (18.17) | 65.1 (17.60) | 65.6 (17.06) | 65.7 (17.62)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 649 | 325 | 646 | 1620
    (all) | 1.6 (0.61) | 1.6 (0.59) | 1.6 (0.64) | 1.6 (0.62)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 18.0 (21.52) | 19.8 (21.51) | 17.9 (22.49) | 18.3 (21.91)
Disease Activity Score 28 Based on CRP (DAS28[CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score ≤ 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 649 | 324 | 647 | 1620
    (all) | 5.8 (0.94) | 5.9 (0.96) | 5.8 (0.97) | 5.8 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: The primary endpoint for United States (US)/Food and Drug Administration (FDA) regulatory purposes was ACR 20% response (ACR20) at Week 12. Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 651 | 327 | 651
percentage of participants | 36.4 [32.7 to 40.1] | 63.0 [57.8 to 68.2] | 70.5 [67.0 to 74.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — In order to preserve Type I error, a step-down approach was used to test the primary and ranked key secondary endpoints in a pre-specified order where statistical significance at the 0.05 level could be claimed for a lower ranked endpoint only if the previous endpoint in the sequence met the requirements of significance; p < 0.001, Cochran-Mantel-Haenszel — This comparison was the primary analysis for US/FDA regulatory purposes, and a ranked key secondary endpoint for EU/EMA regulatory purposes; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 34.1, 95% CI 2-sided [29.0 to 39.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.018, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 7.5, 95% CI 2-sided [1.2 to 13.8] — Response Rate Difference = Upadacitinib - Adalimumab

2. Primary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at Week 12
Description: The primary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes was clinical remission, based on a Disease Activity Score 28 (DAS28)-CRP score of < 2.6 at Week 12.
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 651 | 327 | 651
percentage of participants | 6.1 [4.3 to 8.0] | 18.0 [13.9 to 22.2] | 28.7 [25.2 to 32.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — This comparison was the primary analysis for EU/EMA regulatory purposes, and a ranked key secondary endpoint for US/FDA regulatory purposes; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 22.6, 95% CI 2-sided [18.6 to 26.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 10.7, 95% CI 2-sided [5.3 to 16.1] — Response Rate Difference = Upadacitinib - Adalimumab

3. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Week 12
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at Baseline; multiple imputation was used for missing post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 643 | 319 | 634
units on a scale | -1.15 [-1.276 to -1.017] | -2.01 [-2.175 to -1.848] | -2.48 [-2.608 to -2.347]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for US/FDA and EU/EMA; Analysis of covariance (ANCOVA) model with treatment, prior biological DMARD use, and Baseline value as covariates; LS Mean Difference = -1.33, 95% CI 2-sided [-1.469 to -1.194] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p < 0.001, ANCOVA — This comparison was not part of the pre-specified multiplicity testing sequence; ANCOVA model with treatment, prior biological DMARD use and Baseline value as covariates; LS Mean Difference = -0.47, 95% CI 2-sided [-0.638 to -0.295] — Treatment Difference = Upadacitinib - Adalimumab

4. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 26
Description: The mTSS measures the level of joint damage from radiographs of the hands and feet, assessed by 2 independent, blinded readers. mTSS is calculated as the sum of the total joint erosion score and total joint space narrowing (JSN) score.
  Joint erosion severity was assessed in 16 joints in each hand and wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 280 (worst).
  JSN was assessed in 15 joints of each hand and wrist, and 6 joints of each foot, including subluxation, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 168 (worst).
  The mTSS is the sum of the joint erosion and JSN scores and ranges from 0 (normal) to 448 (worst). A negative change from Baseline in mTSS indicates improvement in joint damage whereas a change from Baseline greater than 0 indicates progression.
Time Frame: Baseline and Week 26
Population: Full analysis set participants with available data at Baseline; linear extrapolation was used for participants who discontinued prior to Week 26 or who were rescued prior to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 599 | 296 | 593
units on a scale | 0.92 [0.64 to 1.20] | 0.10 [-0.25 to 0.46] | 0.24 [-0.04 to 0.53]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; ANCOVA model with treatment, prior biological DMARD use and Baseline value as covariates; LS Mean Difference = -0.67, 95% CI 2-sided [-0.97 to -0.37] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.448, ANCOVA — This comparison was not part of the pre-specified multiplicity testing sequence; ANCOVA model with treatment, prior biological DMARD use and Baseline value as covariates; LS Mean Difference = 0.14, 95% CI 2-sided [-0.23 to 0.51] — Treatment Difference = Upadacitinib - Adalimumab

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 648 | 324 | 644
units on a scale | -0.28 [-0.339 to -0.227] | -0.49 [-0.556 to -0.415] | -0.60 [-0.653 to -0.538]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; ANCOVA model with treatment, prior biological DMARD use and Baseline value as covariates; LS Mean Difference = -0.31, 95% CI 2-sided [-0.372 to -0.253] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.004, ANCOVA — This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for US/FDA only; ANCOVA model with treatment, prior biological DMARD use and Baseline value as covariates; LS Mean Difference = -0.11, 95% CI 2-sided [-0.184 to -0.036] — Treatment Difference = Upadacitinib - Adalimumab

6. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 651 | 327 | 651
percentage of participants | 14.9 [12.2 to 17.6] | 29.1 [24.1 to 34.0] | 45.2 [41.3 to 49.0]
Statistical Analysis 1: Comparison: Adalimumab vs Upadacitinib; Test type: Non-Inferiority — A non-inferiority test of upadacitinib versus adalimumab was evaluated using the lower bound of the 95% confidence interval (CI) of the treatment difference against a non-inferiority margin of 10%. This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for US/FDA only; Response Rate Difference = 16.1, 95% CI 2-sided [9.9 to 22.3] — Response Rate Difference = Upadacitinib - Adalimumab
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for US/FDA only; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 30.3, 95% CI 2-sided [25.6 to 35.0] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 616 | 309 | 616
units on a scale | 3.56 [2.79 to 4.33] | 6.27 [5.31 to 7.23] | 7.89 [7.11 to 8.68]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 3, analysis 1]; MMRM model with fixed effects of treatment, visit, and treatment-by-visit interaction, previous bDMARD use, and Baseline value as covariate; LS Mean Difference = 4.33, 95% CI 2-sided [3.52 to 5.15] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.002, Mixed Effect Model Repeat Measurement — This comparison was not part of the pre-specified multiplicity testing sequence; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = 1.62, 95% CI 2-sided [0.62 to 2.62] — Treatment Difference = Upadacitinib - Adalimumab

8. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12
Description: The DAS28(CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28(CRP) score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 651 | 327 | 651
percentage of participants | 13.8 [11.2 to 16.5] | 28.7 [23.8 to 33.7] | 45.0 [41.2 to 48.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 31.2, 95% CI 2-sided [26.5 to 35.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Non-Inferiority — A non-inferiority test of upadacitinib versus adalimumab was evaluated using the lower bound of the 95% confidence interval (CI) of the treatment difference against a non-inferiority margin of 10%. This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for EU/EMA only; Response Rate Difference = 16.3, 95% CI 2-sided [10.0 to 22.5] — Response Rate Difference = Upadacitinib - Adalimumab
Statistical Analysis 3: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use

9. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity Based on CDAI at Week 12
Description: Low disease activity based on the clinical disease activity index (CDAI) is defined as a CDAI score ≤ 10.
  CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom CDAI data were missing at Week 12 were considered non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 651 | 327 | 651
percentage of participants | 16.3 [13.4 to 19.1] | 30.0 [25.0 to 34.9] | 40.4 [36.6 to 44.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 24.1, 95% CI 2-sided [19.4 to 28.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 10.4, 95% CI 2-sided [4.2 to 16.7] — Response Rate Difference = Upadacitinib - Adalimumab

10. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 12
Description: Participants were asked to indicate the time it took for them to get as limber as possible after awakening with morning stiffness over the past 7 days. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 619 | 306 | 618
minutes | -48.59 [-58.84 to -38.34] | -82.71 [-95.80 to -69.62] | -92.63 [-103.03 to -82.23]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = -44.04, 95% CI 2-sided [-55.39 to -32.69] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.164, Mixed Effect Model Repeat Measurement — This comparison was not part of the pre-specified multiplicity testing sequence; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = -9.92, 95% CI 2-sided [-23.89 to 4.05] — Treatment Difference = Upadacitinib - Adalimumab

11. Secondary Outcome: Change From Baseline in in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: The FACIT Fatigue scale is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a four point Likert scale. The FACIT Fatigue Scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better the quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 613 | 307 | 612
units on a scale | 4.81 [3.85 to 5.77] | 7.44 [6.25 to 8.64] | 8.95 [7.98 to 9.93]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = 4.15, 95% CI 2-sided [3.13 to 5.16] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.017, Mixed Effect Model Repeat Measurement — This comparison was not part of the pre-specified multiplicity testing sequence; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = 1.51, 95% CI 2-sided [0.27 to 2.76] — Treatment Difference = Upadacitinib - Adalimumab

12. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 12
Description: Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100. A score of 0 indicates "no pain" and a score of 100 indicates "worst possible pain." A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 616 | 307 | 614
mm | -15.46 [-17.63 to -13.29] | -25.31 [-28.16 to -22.47] | -31.76 [-33.96 to -29.56]
Statistical Analysis 1: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for US/FDA only; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = -6.45, 95% CI 2-sided [-9.63 to -3.27] — Treatment Difference = Upadacitinib - Adalimumab
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement — This comparison was not part of the pre-specified multiplicity testing sequence; [statistical method as in outcome 7, analysis 1]; LS Mean Difference = -16.30, 95% CI 2-sided [-18.89 to -13.71] — Treatment Difference = Upadacitinib - Placebo

13. Secondary Outcome: Percentage of Participants With No Radiographic Progression at Week 26
Description: No radiographic progression is defined as a change from Baseline in mTSS ≤ 0. The mTSS measures the level of joint damage from radiographs of the hands and feet, which were assessed by 2 independent, blinded readers. mTSS is calculated as the sum of the total joint erosion score and total joint space narrowing (JSN) score and ranges from 0 (normal) to 448 (worst).
  Joint erosion severity was assessed in 16 joints in each hand and wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 280 (worst).
  Joint space narrowing (JSN) was assessed in 15 joints of each hand and wrist, and 6 joints of each foot, including subluxation, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 168 (worst).
Time Frame: Baseline and Week 26
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 599 | 296 | 593
percentage of participants | 76.0 [72.5 to 79.4] | 86.8 [83.0 to 90.7] | 83.5 [80.5 to 86.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — This comparison was a ranked key secondary endpoint in the pre-specified multiplicity testing sequence for EU/EMA only; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 7.5, 95% CI 2-sided [3.0 to 12.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p = 0.187, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = -3.4, 95% CI 2-sided [-8.2 to 1.5] — Response Rate Difference = Upadacitinib - Adalimumab

14. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Adalimumab | Upadacitinib
Number analyzed (Participants) | 651 | 327 | 651
percentage of participants | 4.9 [3.3 to 6.6] | 13.5 [9.8 to 17.2] | 24.9 [21.6 to 28.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 20.0, 95% CI 2-sided [16.3 to 23.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adalimumab vs Upadacitinib; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use; Response Rate Difference = 11.4, 95% CI 2-sided [6.5 to 16.4] — Response Rate Difference = Upadacitinib - Adalimumab

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 26, or up to 30 days after last dose for those receiving placebo or upadacitinib who discontinued prior to Week 26, or up to 70 days after last dose for those receiving adalimumab who discontinued prior to Week 26.
Description: One participant randomized to upadacitinib received placebo to adalimumab but did not receive upadacitinib and is counted in the placebo group for analyses of safety.
  One participant who switched from placebo to upadacitinib at Week 18 did not receive any upadacitinib and is therefore not counted in the placebo / upadacitinib treatment group.
Groups:
- Placebo: Participants received placebo to upadacitinib orally once daily (QD) and placebo to adalimumab by subcutaneous injection once every two weeks (eow) for up to 26 weeks. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 15 mg upadacitinib orally QD.
  Includes events up to the time of rescue (at Weeks 14, 18, 22) or up to Week 26 for those who were not rescued.
- Adalimumab: Participants received placebo to upadacitinib orally QD and 40 mg adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 15 mg upadacitinib orally QD.
  Includes events up to the time of rescue (at Weeks 14, 18, 22) or up to Week 26 for those who were not rescued.
- Upadacitinib: Participants randomized to receive 15 mg upadacitinib orally QD and placebo to adalimumab by subcutaneous injection eow for up to 48 weeks in Period 1. Participants who did not achieve a ≥ 20% improvement in TJC and SJC at Weeks 14, 18, or 22 compared to Baseline were switched to 40 mg adalimumab eow.
  Includes events up to the time of rescue (at Weeks 14, 18, 22) or up to Week 26 for those who were not rescued.
- Placebo / Upadacitinib: Participants who originally received placebo were switched at Weeks 14, 18, or 22 to receive 15 mg upadacitinib orally QD.
  Includes all events that occurred after the switch to rescue treatment up to Week 26.
- Adalimumab / Upadacitinib: Participants who originally received adalimumab were switched at Weeks 14, 18, or 22 to receive 15 mg upadacitinib orally QD.
  Includes all events that occurred after the switch to rescue treatment up to Week 26.
- Upadacitinib / Adalimumab: Participants who originally received 15 mg upadacitinib QD were switched at Weeks 14, 18, or 22 to receive 40 mg adalimumab eow.
  Includes all events that occurred after the switch to rescue treatment up to Week 26.
Arm/Group | Placebo | Adalimumab | Upadacitinib | Placebo / Upadacitinib | Adalimumab / Upadacitinib | Upadacitinib / Adalimumab
All-Cause Mortality (participants affected / at risk) | 2/652 | 2/327 | 0/650 | 0/304 | 0/77 | 0/125
Serious Adverse Events (participants affected / at risk) | 19/652 | 14/327 | 24/650 | 7/304 | 0/77 | 2/125
Other Adverse Events (participants affected / at risk) | 43/652 | 16/327 | 72/650 | 9/304 | 6/77 | 4/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=652) | Adalimumab (N=327) | Upadacitinib (N=650) | Placebo / Upadacitinib (N=304) | Adalimumab / Upadacitinib (N=77) | Upadacitinib / Adalimumab (N=125)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIGHT VENTRICULAR DILATATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRIC POLYPS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALLOPIAN TUBE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INFECTED BITE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIOUS COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AIRWAY COMPLICATION OF ANAESTHESIA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VERTEBRAL LESION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEMYELINATION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROTOXICITY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAPLEGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER PROLAPSE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=652) | Adalimumab (N=327) | Upadacitinib (N=650) | Placebo / Upadacitinib (N=304) | Adalimumab / Upadacitinib (N=77) | Upadacitinib / Adalimumab (N=125)
NASOPHARYNGITIS (Infections and infestations) | 19 (20) | 9 (10) | 36 (42) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 24 (24) | 7 (8) | 37 (43) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02629159/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT02629159/SAP_001.pdf